CLINICAL TRIAL: NCT02124928
Title: Morphological and Serological Criteria of Plaque Vulnerability: Risk Assessment for Symptomatic and Asymptomatic Carotid Artery Stenosis
Acronym: VUCAP
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Prim PD Dr Afshin Assadian (Other)
Collaborators: Wilhelminenspital Vienna (Other)
Responsible Party: Sponsor-Investigator, Prim PD Dr Afshin Assadian, Prim PD Dr, Wilhelminenspital Vienna
Organization: Wilhelminenspital Vienna (Other)
Other Study IDs: VUCAP; EK-11-208-VK (Other: Ethics committee Vienna)
Record Dates: First submitted 2014-04-16; First posted 2014-04-28 (Estimated); Last update posted 2015-09-21 (Estimated); Status verified 2015-09

CONDITIONS: Atherosclerosis; Carotid Artery Disease
Keywords: stroke; biomarkers; vulnerable plaque; carotid endarterectomy; carotid artery disease
MeSH Terms: conditions — Atherosclerosis; Carotid Artery Diseases; Stroke | interventions — Endarterectomy, Carotid

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — whole blood serum carotid artery plaque
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- carotid artery stenosis: Patients with symptomatic or asymptomatic carotid artery stenosis indicated for carotid endarterectomy, who provide written informed consent, will be included in this study. The investigators will compare patients ultrasonographic data, serum laboratory analyses and histomorphological preferances to look for biomarkers for the plaque instability.
  Interventions: Procedure: Carotid endarterectomy

INTERVENTIONS:
Procedure: Carotid endarterectomy — Carotid endarterectomy is a surgery used to reduce the risk of stroke, by correcting stenosis in the carotid artery. Endarterectomy is the removal of material on the inside (end-) of an artery.An incision is made on the midline side of the Sternocleidomastoid muscle. The incision is between 5 and 10 cm in length. Then the patients get 5000 IU heparin by the anesthesia. The internal, common and external carotid arteries are carefully identified, controlled with vessel loops, and clamped. The lumen of the internal carotid artery is opened, and the atheromatous plaque removed. The artery is closed using suture. The procedure is performed under local anesthesia. Local anesthesia, opposite to general, allows for direct monitoring of neurological status by intra-operative verbal contact and testing of grip strength.

SUMMARY:
The aim of this study is to investigate the association of sonographic and histological features of the plaque among each other and with biomarkers of cardiovascular risk. The predictive value of these factors concerning the long-term clinical outcome after carotid endarterectomy will also be assessed. This may help to improve the identification of patients with carotid artery stenosis who will benefit most from carotid endarterectomy. The investigators major hypothesis is that the morphology of carotid plaques is associated with objectifiable sonographic parameters, in particular with the greyscale median. Second, the investigators hypothesize that sonographic and histological plaque morphology are associated with certain biomarkers of cardiovascular risk. Identification of 'vulnerable plaques' on the basis of a peripheral blood draw and a sonographic investigation may enable the treating physician to focus resources on patients who will benefit most form therapeutic interventions for primary prevention of ischemic stroke.

DETAILED DESCRIPTION:
The indication for revascularization of carotid artery stenoses is typically based on the degree of stenosis and the presence of symptoms. Recent evidence suggests that the risk of embolization from an atherosclerotic plaque may be associated with plaque density as assessed sonographically by determination of the greyscale median. Also, an association of serum proteins vascular endothelial growth factor (VEGF), hypoxia inducible factor (HIF) and pigment epithelium-derived factor (PEDF), matrix metalloproteinases 2, 8 and 9 with unstable plaques has been reported.

The VUCAP study will include patients undergoing carotid endarterectomy for symptomatic or asymptomatic carotid artery disease. Sonographic and serological markers of plaque vulnerability will be compared with histological features of the plaque and clinical presentation (symptomatic vs. asymptomatic). Preoperatively, the greyscale median of the plaque is assessed. Histomorphological investigation of the carotid plaques will be performed. Serological investigations will include markers of inflammation, thrombo-modulatory factors, lipid fractions and other parameters that have been associated with unstable plaques.

The aim of the present study is to assess the ability of pigment epithelium-derived factor (PEDF), vascular endothelial growth factor (VEGF), hypoxia-induced factor 1 alpha (HIF 1-α), matrix metalloproteinases 2, 8 and 9 to differentiate between vulnerable and stable carotid artery plaques. Identification of 'vulnerable plaques' on the basis of a peripheral blood draw and a sonographic investigation may enable the treating physician to focus resources on patients who will benefit most form therapeutic interventions for primary prevention of ischemic stroke.

ELIGIBILITY:
Inclusion Criteria:

* asymptomatic stenosis of internal carotid artery >70%
* symptomatic stenosis of internal carotid artery >60%
* planed surgical treatment of the stenosis

Exclusion Criteria:

* pregnancy
* symptomatic coronary heart disease
* myocardial infarction or acute coronary syndrome in the past 3 months
* acute peripheral artery occlusion in the past 3 months
* immaturity
* existence of a guardianship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Four hundred patients with symptomatic or asymptomatic carotid artery stenosis undergoing carotid endarterectomy, after written informed consent will be included in this study. The inclusion would be done through our ambulatory care clinic.
Sampling Method: Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2012-09; Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
serum levels of PEDF, VEGF, HIF-1 alpha, MMP-2, -8 and -9 compared to histomorphological classification of the plaque based on AHA classification and ultrasonographic data- grey scale median (GSM) | ultrasonographical data are assessed a day before the surgery, carotid artery plaque will be taken during the surgery, whole blood on the day of operation,
  Extended sonomorphological investigation will be performed by a sonographer blinded to patients' characteristics, for the assessment of grey scale median (GSM). After removal plaques will be fixated in RNAlater for further RNA-determinations. In addition, histomorphological characterization of the plaque will be performed and the plaque classified based on the American Heart Association (AHA) classification. RNA-determination will focus on the expression levels of PEDF. VEGF, HIF-1 alpha, MMP-2, -8 and -9. For that purpose we will perform RNA isolation from the tissue, transcription to cDNA and also a quantitative real-time PCR. Furthermore immunostaining of the plaque with PEDF, VEGF, HIF-1 alpha, MMP-2, -8 and -9 antibodies to determine the distribution of those proteins within the plaques will be done.

SECONDARY OUTCOMES:
change in blood serum levels as well as protein level expression of PEDF, VEGF, HIF-1 alpha, MMP-2, -8 and -9 after plaque removal | serum blood levels are evaluated from the whole blood twice: on the day of surgery and 6 weeks after removal of the plaque
  enzyme-linked immunosorbent assay (ELISA) will be done for the determination of PEDF, VEGF, HIF-1 alpha, before and after surgery

OTHER OUTCOMES:
composite end point of death, stroke, myocardial infarction | From date of randomization until the date of first documented or date of death from any cause assessed up to 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Afshin Assadian, Prim PD Dr, Principal Investigator — Georg Hagmüller Institute for Vascular Research Wilheminenspital Vienna, Austria
Locations (1):
- Surgery Departement, Georg Hagmüller Institute for Vascular Research Wilheminenspital, Vienna, Austria